CLINICAL TRIAL: NCT06143904
Title: An Open-Label Study to Evaluate the Absolute Bioavailability of Genz-112638 and the Absorption, Metabolism, and Excretion of [14C]-Genz-112638 in Male Subjects
Brief Title: A Study to Evaluate Absolute Bioavailability, Absorption, Metabolism, and Excretion of Genz-112638 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: GZGD02107; U1111-1294-7994 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Gaucher's Disease Type I
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Period 1 -2 (Experimental): Single-dose Intravenous (IV) Genz-112638 Day 1 followed by single dose GenZ-112638 oral capsules Day 8
  Interventions: Drug: Genz-112638
- Treatment Period 1-4 (Experimental): Single-dose Intravenous (IV) Genz-112638 Day 1; single dose GenZ-112638 oral capsules Day 8; oral capsule Genz-112638 Days 9-14; single dose [14C]-Genz-112638 oral solution Day 15
  Interventions: Drug: Genz-112638; Drug: [14C]-Genz-112638

INTERVENTIONS:
Drug: Genz-112638 — Pharmaceutical form:Solution-Route of administration:IV
  Other Names: GZ385660/ eliglustat; Cerdelga
Drug: Genz-112638 — Pharmaceutical form:Capsule-Route of administration:Oral
  Other Names: GZ385660/ eliglustat
Drug: [14C]-Genz-112638 — Pharmaceutical form:Solution-Route of administration:Oral
  Other Names: GZ385660/ eliglustat
  Arms: Treatment Period 1-4

SUMMARY:
Objectives:

To determine pharmacokinetic (PK) variables, including absolute bioavailability (F), of Genz-99067, the free base of the L-tartaric acid salt of Genz-112638 as it exists in plasma, after a single intravenous (IV) dose and after a single oral dose of Genz-112638 (unlabeled).

To determine the PK, total recovery, routes and rates of excretion, and the metabolic profile of Genz-99067 after 5 days of BID oral dosing with unlabeled Genz-112638 followed by a single dose of [14C]-Genz-112638.

DETAILED DESCRIPTION:
The maximum study duration for an individual subject was approximately 65 days from the beginning of Screening through the Safety Follow-up visit.

ELIGIBILITY:
Inclusion Criteria: Having given written informed consent prior to undertaking any study-related procedure The subject has a body weight of 50 to 100 kg [110 to 220 pounds (lb)] with a body mass index (BMI) less than 30 kilograms per square meter (kg/m2) at Screening.

The subject's physical examination results, vital signs, laboratory assessments, and cardiac assessments are within normal limits or, if abnormal, are not clinically significant at Screening and Day -1. Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

Prolonged QTc interval (eg, repeated demonstration of a QTc interval ≥450 msec), family history of long QT or Brugada Syndrome, and/or history of sudden death in a first-degree relative.

The subject receives an immunization within 30 days of providing informed consent.

The subject has a history of drug allergies (eg, significant rash, hives, etc in response to antibiotics).

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06-03 (Actual); Primary Completion 2009-07-05 (Actual); Study Completion 2009-07-05 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetic (PK) parameter: Cmax | Multiple timepoints up to Day 26
  Plasma concentrations of Genz-99067 will be collected at pre-specified timepoints
Assessment of pharmacokinetic (PK) parameter: Tmax | Multiple timepoints up to Day 26
  Plasma concentrations of Genz-99067 will be collected at pre-specified timepoints
Assessment of pharmacokinetic (PK) parameter: AUC0-∞ | Multiple timepoints up to Day 26
  Plasma concentrations of Genz-99067 will be collected at pre-specified timepoints
Assessment of pharmacokinetic (PK) parameter: AUC0 -τ | Multiple timepoints up to Day 26
  Plasma concentrations of Genz-99067 will be collected at pre-specified timepoints
Assessment of pharmacokinetic (PK) parameter: AUC0-∞/D | Multiple timepoints up to Day 26
  Plasma concentrations of Genz-99067 will be collected at pre-specified timepoints
Assessment of pharmacokinetic (PK) parameter: AUC0-τ/D | Multiple timepoints up to Day 26
  Plasma concentrations of Genz-99067 will be collected at pre-specified timepoints
Assessment of pharmacokinetic (PK) parameter: F | Multiple timepoints up to Day 26
  Plasma concentrations of Genz-99067 will be collected at pre-specified timepoints
Assessment of pharmacokinetic (PK) parameter: CL/F | Multiple timepoints up to Day 26
  Plasma concentrations of Genz-99067 will be collected at pre-specified timepoints
Assessment of pharmacokinetic (PK) parameter: t½ | Multiple timepoints up to Day 26
  Plasma concentrations of Genz-99067 will be collected at pre-specified timepoints
Pharmacokinetic (PK) parameter: Absolute bioavailability (F) of single-dose oral versus single-dose IV administration | Multiple timepoints up to Day 26
Assessment of pharmacokinetic (PK) parameter: Total radioactivity excreted in urine and feces | Multiple timepoints up to Day 26
  Total radioactivity excreted in urine and feces will be converted to percentage of radioactive dose.
Assessment of pharmacokinetic (PK) parameter: Total radioactivity in whole blood and plasma | Multiple timepoints up to Day 26
  Total radioactivity in whole blood and plasma will be converted to ngEq/g Genz-99067 concentration for whole blood and ngEq/mL for plasma, based on the dose specific activity.
Assessment of pharmacokinetic (PK) parameter: % relative abundance of each component in samples of plasma or excreta | Multiple timepoints up to Day 26
  It will be estimated as [(radioactivity for the HPLC peak)/(total radioactivity injected per HPLC run) x 100].
Assessment of pharmacokinetic (PK) parameter: The percentage of the administered dose attributed to each component in samples of urine or feces | Multiple timepoints up to Day 26
  It will be estimated as [(% relative abundance)/100 x (percentage of radioactive dose in the sample)].
Assessment of pharmacokinetic (PK) parameter: The radioactivity of [14C]-Genz-99067 and each major metabolite in plasma, as identified by radio-profiling | Multiple timepoints up to Day 26
  It will be converted to equivalent concentrations as [(% relative abundance)/100 x (equivalent concentration of total radioactivity in the sample)].
Noncompartmental PK parameters: AUC0-t | Multiple timepoints up to Day 26
Noncompartmental PK parameters: AUC0-∞ | Multiple timepoints up to Day 26
Noncompartmental PK parameters: Cmax | Multiple timepoints up to Day 26
Noncompartmental PK parameters: Tmax | Multiple timepoints up to Day 26
Noncompartmental PK parameters: t½ | Multiple timepoints up to Day 26
Noncompartmental PK parameters: Vz/F | Multiple timepoints up to Day 26
Noncompartmental PK parameters: CL/F | Multiple timepoints up to Day 26
Noncompartmental PK parameters for urine and feces: Cum Ae | Multiple timepoints up to Day 26
Noncompartmental PK parameters for urine and feces: % dose | Multiple timepoints up to Day 26
Renal clearance (CLR) for total plasma radioactivity and Genz-99067 | Multiple timepoints up to Day 26
PK parameters [AUC0-τ, AUC0-∞, Cmax, Tmax, t½] and metabolite ratio for metabolite(s) of Genz-99067 | Multiple timepoints up to Day 26

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs), serious adverse event (SAEs), and adverse event of special interest (AESI) | Up to Day 33

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org